CLINICAL TRIAL: NCT03500731
Title: Lung Transplant in Tandem With Bone Marrow Transplant for Combined Lung and Bone Marrow Failure
Brief Title: Lung and Bone Marrow Transplantation for Lung and Bone Marrow Failure
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Paul Szabolcs (Other)
Responsible Party: Sponsor-Investigator, Paul Szabolcs, Chief, Division of Blood and Marrow Transplantation and Cellular Therapy, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19110120
Record Dates: First submitted 2018-03-30; First posted 2018-04-18 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Idiopathic Pulmonary Fibrosis; Emphysema or COPD
Keywords: Lung Transplantation; Stem Cell Transplantation; Idiopathic Pulmonary Fibrosis; Emphysema or COPD; Bone marrow transplantation; Cadaveric donor; Unrelated donor; HLA-Mismatch; BMT; HSCT; IPF; Pulmonary fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Emphysema; Pulmonary Disease, Chronic Obstructive; Pulmonary Fibrosis | interventions — Rituximab; Alemtuzumab; fludarabine; fludarabine phosphate; Thiotepa; Granulocyte Colony-Stimulating Factor; Filgrastim; Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lung and Bone Marrow Transplantation (Experimental): All patients will undergo a cadaveric, partially HLA-matched lung transplantation followed by a CD3+/CD19+ depleted BMT from the same donor. In this study, the investigators will use a ≥1/6 HLA-matched T cell depleted bone marrow transplantation from a cadaveric organ donor with an identical ABO blood type as the recipient. Prior to transplantation, the marrow will be negatively selected for CD3/CD19 using a CliniMACS® depletion device.
  Subjects will undergo lung transplantation utilizing standard induction regimens selected by the CO-PIs based on the subject's underlying comorbidities and allosensitization. Rituximab may be initiated prior to the lung transplantation with tacrolimus as the ongoing maintenance immunosuppression.
  Subjects will undergo BMT utilizing CD3+/CD19+-depleted bone marrow with bone marrow conditioning beginning no less than 8 weeks after lung transplantation. Bone marrow will be recovered alongside solid organs and will be processed and cryopreserved.
  Interventions: Biological: CD3/CD19 negative hematopoietic stem cells; Drug: Rituximab; Drug: Alemtuzumab; Drug: Fludarabine; Drug: Thiotepa; Drug: G-CSF; Drug: Hydroxyurea

INTERVENTIONS:
Biological: CD3/CD19 negative hematopoietic stem cells — Negative selection for CD3/CD19 will be performed on CliniMACS® depletion device and given at time no less than 8 weeks post lung transplantation
Drug: Rituximab — Transplantation Conditioning
  Other Names: Rituxan
Drug: Alemtuzumab — Transplantation Conditioning
  Other Names: Campath-1H
Drug: Fludarabine — Transplantation Conditioning
  Other Names: Fludara, Oforta
Drug: Thiotepa — Transplantation Conditioning
Drug: G-CSF — Transplantation conditioning
  Other Names: Neupogen, Granix, Zarxio, Filgrastim
Drug: Hydroxyurea — Transplantation Conditioning

SUMMARY:
The purpose of this study is to determine whether a lung transplantation prior to bone marrow transplantation (BMT) would allow for restoration of pulmonary function prior to BMT, allowing to proceed to BMT, to restore hematologic function.

DETAILED DESCRIPTION:
The primary purpose of the study is to evaluate the safety and efficacy of performing lung transplantation followed by cadaveric, partially HLA-matched (≥1/6 HLA-match with an identical ABO blood type) CD3+/CD19+ depleted bone marrow transplantation in bone marrow failure and end-stage lung disease. Idiopathic pulmonary fibrosis (IPF) is a chronic, progressive, and fatal interstitial lung disease for which lung transplantation is the only therapy shown to prolong survival. Given the association of IPF with hematologic cytopenias and bone marrow failure, it is proposed that a tandem lung transplantation and bone marrow transplantation from a single cadaveric donor could be successful. This protocol focuses on performing combined transplantation for candidates that are unable to undergo standard lung transplantation. Lung transplantation prior to bone marrow transplantation (BMT) would allow for restoration of pulmonary function prior to BMT, and to restore hematologic function post BMT transplantation. The secondary objectives are to evaluate the feasibility and long-term complications associated with combined solid organ and BMT including the ability to initiate and successfully withdraw from immunosuppression following BMT and to attain independence from growth factors, red blood cell or platelet transfusions.

ELIGIBILITY:
Inclusion Criteria:

Individuals must meet all of the following criteria in order to be eligible for this study.

1. Subject must be able to understand and provide informed consent.
2. Male or female, 18 through 60 years old, inclusive, at the time of informed consent.
3. Meet criteria for UNOS listing for lung transplantation.
4. Patients must have evidence of end stage lung disease. Examples of such diseases include but are not limited to:

   * Pulmonary Fibrosis
   * COPD/Emphysema
5. Patients must have evidence of bone marrow failure with abnormal low cell count in at least one hematopoietic line, making the patient a poor candidate for long-term immunosuppressive therapy. Eligible patients must meet at least one of the following criteria:

   * Unexplained, non-drug induced neutropenia with absolute neutrophils counts of <1500/µL the previous year, confirmed by repeat testing
   * Unexplained, non-drug induced thrombocytopenia with mean platelets counts of <100,000/µL the previous year, confirmed by repeat testing
   * Unexplained, non-hemolytic anemia, with a hemoglobin level of < 12 g/dL the previous year, confirmed by repeat testing
6. GFR ≥45 mL/min/1.73 m2.
7. AST, ALT ≤4x upper limit of normal, total bilirubin ≤ 2.5 mg/dL, normal INR, albumin >3.0 g/dL
8. Cardiac ejection fraction ≥ 40% or shortening fraction ≥26%.
9. Negative pregnancy test for females, unless surgically sterilized.
10. All females of childbearing potential and sexually active males must agree to use a FDA approved method of birth control for up to 24 months after BMT or for as long as they are taking any medication that may harm a pregnancy, an unborn child or may cause birth defect.
11. Subject will also be counseled regarding the potential risks of infertility following BMT and advised to discuss sperm banking or oocyte harvesting.

Exclusion Criteria:

Individuals who meet any of these criteria are not eligible for this study.

1. Inability or unwillingness of a participant to give written informed consent or comply with study protocol.
2. Patients who have underlying malignant conditions.
3. Patients who have non-malignant conditions not requiring BMT.
4. HIV positive by serology or PCR, HTLV positive by serology. If HTLV serology is positive, it will be confirmed by nucleic acid testing (NAT). If HTLV NAT is negative, subject will remain eligible regardless of HTLV serology result.
5. Females who are pregnant or who are lactating.
6. Allergy to DMSO or any other ingredient used in the manufacturing of the stem cell product.
7. Uncontrolled pulmonary infection, as determined by radiographic findings and/or significant clinical deterioration. NOTE: Pulmonary colonization with multiple organisms is common and will not be considered an exclusion criterion.
8. Uncontrolled infection, as determined by the appropriate imaging and/or confirmatory testing e.g. blood cultures, PCR testing, etc.
9. Recent recipient of any licensed or investigational live attenuated vaccine(s) within 4 weeks of transplant.
10. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2018-04-19 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Death | Up to 2 years post stem cell transplant
  How many, if any, patients die
Engraftment failure | Up to 2 years post stem cell transplant
  How many, if any, develop engraftment failure
Non-hematologic events | Up to 2 years post stem cell transplant
  Any Grade 4 event that happens at any time points
Hematological events | after 30 days post stem cell transplant
  Any Grade 4 hematological events
BOS Score | at 1 year post lung transplant
  Bronchiolitis Obliterans Syndrome (BOS) score based off patient pulmonary function testing. Graded on scale (BOS0 to BOS3), BOS0 having a better outcome then BOS3
T-cell Chimerism | at 12 months post stem cell transplant
  The number of patients who have ≥25% donor T-cell chimerism
Myeloid chimerism | at 12 months post stem cell transplant
  The number of patients with myeloid disorders who attain ≥ 10% myeloid chimerism
Restoration of blood cell count (in absence of growth factors) | at 12 months post stem cell transplant
  Absolute neutrophil count (ANC)≥1000 per microliter of blood, platelets ≥50000 per microliter of blood and hematocrit ≥8 grams per deciliter of blood

SECONDARY OUTCOMES:
Feasibility of patients able to proceed to BMT within 6 months following lung transplantation | Up to 2 years post stem cell transplant
  The number of patients who are able to proceed to BMT within 6 months following lung transplantation
Independence | up to 2 years post stem cell transplant
  The number of patients who are able to be independent from transfusions and growth factors for at least 7 days
Independence | Up to 2 years post stem cell transplant
  The number of patients who are able to be independent from transfusions and growth factors for at least 1 month
Tolerance development to both host and pulmonary grafting | Up to 2 years post stem cell transplant
  Development of tolerance to both the host and pulmonary graft
Long-term complications | Up to 2 years post stem cell transplant
  Long-term complications of combined solid organ and BMT
Acute cellular rejection | Up to 2 years post stem cell transplant
  The number of patients who develop acute cellular rejection
Acute graft-versus-host-disease (GVHD) | Up to 2 years post stem cell transplant
  The number of patients who develop acute graft-versus-host-disease (GVHD)
Chronic graft-versus-host-disease (GVHD) | Up to 2 years post stem cell transplant
  The number of patients who develop chronic graft-versus-host-disease (GVHD)
Ability to withdrawal immunosuppression | By 1 year post stem cell transplant
  The number of patients who are able to start immunosuppression withdrawal.
Time to withdraw immunosuppression | Up to 2 years post stem cell transplant
  Time from BMT to withdrawal of immunosuppression
Prophylactic antimicrobial drugs | Up to 2 years post stem cell transplant
  Time from BMT to independence for prophylactic antimicrobial drugs
Treatment antimicrobial drugs | up to 2 years post stem cell transplant
  Time from BMT to independence from treatment antimicrobial drugs
Chronic lung allograft dysfunction | 1 year post lung transplant
  The number of patients who develop chronic lung allograft dysfunction post lung transplant for all subjects, lung only and lung +stem cell transplant.

OTHER OUTCOMES:
Pace of immune reconstitution | Up to 2 years post stem cell transplant
  The pace of immune reconstitution, systemically and in mucosal surfaces
Mixed chimerism | at Months 1, 3, 6 and 12 post stem cell transplant
  The number of patients who have the incidence of mixed chimerism (.5% host cells)
In vitro immune tolerance | Up to 2 years post stem cell transplant
  The number of patients who have in vitro immune tolerance

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - UPMC Presbyterian, Pittsburgh, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No